CLINICAL TRIAL: NCT07213869
Title: Study of Personalized Alpha tACS for the Recovery of Disorders of Consciousness : Controlled Evaluation With a Single Case Experimental Design
Brief Title: Alpha tACS for Disorders of Consciousness : a Single Case Experimental Design
Acronym: SPARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL24_0976; 2025-A02086-43 (Other: ID-RCB)
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Disorder of Consciousness
Keywords: disorders of consciousness; tACS; tES; transcranial electric stimulation; traumatic brain injury
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Single-Case Experimental Design (SCED, A-B-A-B-A-B): Each participant serves as their own control and undergoes six consecutive phases over approximately three months, alternating between baseline (no stimulation) and active stimulation periods (two weeks each). This intra-subject design maximizes sensitivity to individual changes while limiting confounding from clinical heterogeneity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpha tACS (Experimental): Participants receive Alpha tACS daily, in repeated sessions delivered during three 2-week stimulation periods, alternating with three 2-week no-stimulation (baseline) periods, for a total duration of approximately three months.
  Interventions: Device: Transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: Transcranial alternating current stimulation (tACS) — Alpha tACS daily, in repeated sessions delivered during three 2-week stimulation periods, alternating with three 2-week no-stimulation (baseline) periods, for a total duration of approximately three months

SUMMARY:
BRIEF SUMMARY * (Include a statement of the study hypothesis) Avoid all personal pronouns (Limit: 5000 characters) Disorders of consciousness (DoC) following a severe traumatic brain injury represent a major medical challenge, with very limited therapeutic options and many patients remaining in a minimally conscious state or vegetative/unresponsive wakefulness state for months. To date, only two pharmacological treatments (amantadine and zolpidem) have shown partial benefits. Non-invasive neuromodulation techniques such as transcranial direct current stimulation (tDCS) have produced modest but encouraging results.

Recent advances in transcranial alternating current stimulation (tACS) have demonstrated its ability to modulate brain oscillations, particularly in the alpha frequency range (8-12 Hz), which plays a central role in large-scale functional connectivity, especially within the default mode network (DMN). Neuroimaging studies suggest alpha activity and DMN connectivity are major correlate of the level of consciousness in DoC. Yet experimental evidence suggests that alpha tACS can enhance alpha power and antero-posterior connectivity in healthy subjects, as well as connectivity within the default mode network (DMN). However, no controlled study has yet evaluated its therapeutic potential in patients with DoC.

The present study (SPARC) is a single-center clinical investigation aiming to assess the clinical efficacy of alpha tACS in patients with DoC after traumatic brain injury. The primary hypothesis is that repeated sessions of alpha tACS will improve the level of consciousness, compared to baseline and non-stimulation periods, by reinforcing power and functional connectivity in the alpha band.

This trial adopts a Single-Case Experimental Design (SCED), a robust methodology particularly suited to rare and heterogeneous clinical populations such as DoC. Five adult patients (aged 18-70 years) with DoC persisting for 3-12 months post-trauma will be included. Each participant will undergo six consecutive phases over three months: three non-stimulation (baseline/washout) periods and three stimulation periods, each period lasting two weeks, in an A-B-A-B-A-B sequence. This intra-subject design allows each patient to serve as their own control, maximizing sensitivity to individual changes and limiting confounding by clinical heterogeneity.

The primary outcome measure is the change in the Simplified Evaluation of Consciousness Disorders (SECONDS) score, a validated clinical scale routinely used in DoC assessment. SECONDS will be measured three times weekly throughout the study. Secondary outcomes include: (1) EEG-based classification of consciousness state using an established machine-learning algorithm, (2) spectral power and functional connectivity changes in the alpha band, and (3) resting-state fMRI measures of DMN connectivity. These multimodal assessments aim both to provide objective evidence of clinical improvement and to explore the underlying neurophysiological mechanisms of tACS.

Safety and tolerability are monitored. Previous studies confirm that tACS is safe and well-tolerated, with only minor, transient side effects (tingling, scalp redness, phosphene perception). The study also involves EEG and MRI recordings, both of which are non-invasive and carry only minimal risks.

This study, although limited to five patients, is designed to provide rigorous individual-level evidence of efficacy and mechanistic plausibility. If results demonstrate consistent clinical and neurophysiological improvements, they will justify the design of a larger confirmatory trial and contribute to the development of novel therapeutic approaches for this severely disabled population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Persistent disorder of consciousness (vegetative state/unresponsive wakefulness syndrome or minimally conscious state) according to the Coma Recovery Scale-Revised (CRS-R), lasting 3 to 12 months after traumatic brain injury at the time of the inclusion
* No evidence of exit from minimally conscious state (eMCS) according to Coma Recovery Scale-Revised (CRS-R)

Exclusion Criteria:

* Active epilepsy or major pre-existing central nervous system disorders

  * Craniectomy without bone flap replacement, non-healed scalp lesions, intracerebral metallic implants (except titanium), or implanted electronic devices (e.g., pacemaker)
  * Contraindications to MRI (non-compatible devices, metallic fragments, recent tattoos, etc.)
  * Pregnant or breastfeeding women
  * Persons deprived of liberty, under psychiatric care, or not affiliated with a social security/health insurance system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in SECONDS score (Simplified Evaluation of CONsciousness Disorders) during tACS vs. non-stimulation phases | Assessed 3 times per week throughout the 12-week protocol (across six phases: three stimulation and three non-stimulation periods).
  The primary endpoint is the evolution of the SECONDS score, a standardized and validated clinical scale (range 1-8) routinely used in disorders of consciousness.
  Each participant is analyzed individually (single-case time series). Scores during three active stimulation phases will be compared with scores during three non-stimulation phases.

SECONDARY OUTCOMES:
EEG-based classification of consciousness state (SVM algorithm) | Baseline and end of each stimulation and non-stimulation phase (8 EEG recordings per participant over 12 weeks, plus 1-month follow-up).
  Change in the EEG-derived classification score using a validated support vector machine algorithm (Sitt et al. 2014), which estimates probability of being in vegetative state vs. minimally conscious state.
  Each participant is analyzed individually (single-case time series). We will compare the variation of this score between stimulation and non-stimulation phases.
Change in alpha spectral power and antero-posterior functional connectivity (EEG) | Baseline and end of each stimulation and non-stimulation phase (8 EEG recordings per participant over 12 weeks, plus 1-month follow-up).
  Evolution of alpha-band (8-12 Hz) spectral power and antero-posterior functional connectivity measured by EEG, analyzed for changes between stimulation and non-stimulation periods.
  Each participant is analyzed individually (single-case time series).
Resting-state fMRI connectivity within the Default Mode Network (DMN) | At study start, after 2 weeks without stimulation, and after 2 weeks of stimulation (3 MRI scans per participant).
  Change in functional connectivity within the default mode network (seed-based resting-state fMRI analysis) between baseline, post-non-stimulation, and post-stimulation phases, and association with clinical response to tACS.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline HERAULT, Dr, Study Chair — Hospices Civils de Lyon
Locations (1):
- Post-Intensive Care Neurorehabilitation Unit (Service de Reeducation Post-Reanimation) in Pierre Wertheimer Neurologic Hospital, Bron, France

IPD SHARING:
Plan to Share IPD: No